CLINICAL TRIAL: NCT00005970
Title: Phase III Trial of Doxorubicin and Cyclophosphamide (AC) Followed by Weekly Paclitaxel With or Without Trastuzumab as Adjuvant Treatment for Women With HER-2 Over-Expressing or Amplified Node Positive or High-Risk Node Negative Breast Cancer
Brief Title: Doxorubicin Hydrochloride, Cyclophosphamide, and Pacltaxel With or Without Trastuzumab in Treating Women With HER2-Positive Node-Positive or High-Risk Node-Negative Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Cancer and Leukemia Group B (Network); Eastern Cooperative Oncology Group (Network); Canadian Cancer Trials Group (Network); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01849; NCI-2012-01849 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9343; ECOG-N9831; CAN-NCIC-MA28; SWOG-N9831; MA.28; NCCTG-N9831; CALGB-49909; CDR0000067953; GUMC-00224; N9831 (Other: Alliance for Clinical Trials in Oncology); N9831 (Other: CTEP); U10CA180821 (NIH); U10CA025224 (NIH)
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Breast Adenocarcinoma; HER2 Positive Breast Carcinoma; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage IIIA Breast Cancer AJCC v7
MeSH Terms: conditions — Breast Neoplasms | interventions — Aromatase Inhibitors; Cyclophosphamide; Doxorubicin; Paclitaxel; Taxes; Tamoxifen; Trastuzumab; PF-05280014; Ogivri; Ontruzant; trastuzumab biosimilar HLX02

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (AC, paclitaxel, tamoxifen, aromatase inhibitor) (Experimental): Patients receive doxorubicin hydrochloride IV and cyclophosphamide IV over 20-30 minutes on day 1. Treatment repeats every 3 weeks for 4 courses. Patients then receive paclitaxel IV over 1 hour beginning on day 1 of week 13 and continuing weekly for 12 courses in the absence of disease progression or unacceptable toxicity. Within 5 weeks after completion of paclitaxel, patients may undergo radiotherapy. All postmenopausal ER- or PR-positive patients receive oral tamoxifen or an aromatase inhibitor once daily for 5 years beginning no later than 5 weeks after the last dose of paclitaxel. Patients may also receive an aromatase inhibitor once daily for 5 years after 5 years of daily tamoxifen. Patients who receive tamoxifen once daily for less than 4.5 years may receive an aromatase inhibitor daily until they have received a total of 5 years of adjuvant hormonal therapy.
  Interventions: Drug: Aromatase Inhibition Therapy; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Tamoxifen Citrate
- Arm II (AC, paclitaxel, trastuzumab, tamoxifen) (Experimental): Patients receive doxorubicin hydrochloride, cyclophosphamide, and paclitaxel as in arm I. Patients then receive trastuzumab (Herceptin®) IV over 30-90 minutes beginning on day 1 of week 25 and continuing weekly for 52 courses in the absence of disease progression or unacceptable toxicity. Within 5 weeks after completion of paclitaxel, patients may undergo radiotherapy. All postmenopausal ER- or PR-positive patients receive oral tamoxifen or an aromatase inhibitor once daily for 5 years beginning no later than 5 weeks after the last dose of paclitaxel. Patients may also receive an aromatase inhibitor once daily for 5 years after 5 years of daily tamoxifen. Patients who receive tamoxifen once daily for less than 4.5 years may receive an aromatase inhibitor daily until they have received a total of 5 years of adjuvant hormonal therapy.
  Interventions: Drug: Aromatase Inhibition Therapy; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Tamoxifen Citrate; Biological: Trastuzumab
- Arm III (AC, paclitaxel, trastuzumab, tamoxifen) (Experimental): Patients receive doxorubicin hydrochloride and cyclophosphamide as in arm I. Patients then receive paclitaxel IV over 1 hour and trastuzumab IV over 30-90 minutes beginning on day 1 of week 13 and continuing weekly for 12 courses. Patients then receive trastuzumab IV over 30 minutes beginning on day 1 of week 25 and continuing weekly for 40 courses in the absence of disease progression or unacceptable toxicity.
  Within 5 weeks after completion of paclitaxel, patients may undergo radiotherapy. All postmenopausal ER- or PR-positive patients receive oral tamoxifen or an aromatase inhibitor once daily for 5 years beginning no later than 5 weeks after the last dose of paclitaxel. Patients may also receive an aromatase inhibitor once daily for 5 years after 5 years of daily tamoxifen. Patients who receive tamoxifen once daily for less than 4.5 years may receive an aromatase inhibitor daily until they have received a total of 5 years of adjuvant hormonal therapy.
  Interventions: Drug: Aromatase Inhibition Therapy; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Tamoxifen Citrate; Biological: Trastuzumab

INTERVENTIONS:
Drug: Aromatase Inhibition Therapy — Given orally
  Other Names: Aromatase Inhibition
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Tamoxifen Citrate — Given orally
  Other Names: Apo-Tamox; Clonoxifen; Dignotamoxi; Ebefen; Emblon; Estroxyn; Fentamox; Gen-Tamoxifen; Genox; ICI 46,474; ICI-46474; Jenoxifen; Kessar; Ledertam; Lesporene; Nolgen; Noltam; Nolvadex; Nolvadex-D; Nourytam; Novo-Tamoxifen; Novofen; Noxitem; Oestrifen; Oncotam; PMS-Tamoxifen; Soltamox; TAM; Tamax; Tamaxin; Tamifen; Tamizam; Tamofen; Tamoxasta; Tamoxifeni Citras; Zemide
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; ALT02; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Herzuma; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; Ogivri; Ontruzant; PF-05280014; rhuMAb HER2; RO0452317; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab-dkst; Trastuzumab-DTTB; Trastuzumab-pkrb; Trastuzumab-QYYP; Trazimera
  Arms: Arm II (AC, paclitaxel, trastuzumab, tamoxifen); Arm III (AC, paclitaxel, trastuzumab, tamoxifen)

SUMMARY:
This randomized phase III trial studies doxorubicin hydrochloride, cyclophosphamide, paclitaxel, and trastuzumab to see how well they work compared to combination chemotherapy alone in treating women with breast cancer that is human epidermal growth factor receptor 2 (HER2)-positive and has spread to the lymph nodes or high-risk and has not spread to the lymph nodes. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. It is not yet known whether combination chemotherapy is more effective with or without trastuzumab in treating breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the combination of doxorubicin hydrochloride and cyclophosphamide (AC) followed by weekly paclitaxel with the combination of AC followed by the combination of weekly paclitaxel and trastuzumab in terms of disease free survival (DFS). (Stage I) II. To compare the combination of AC followed by weekly paclitaxel with the combination of AC followed by the combination of weekly paclitaxel and trastuzumab in terms of the rate of cardiac events. (Stage I) III. To compare the combination AC followed by weekly paclitaxel with the sequential schedule of the combination of AC, weekly paclitaxel, and trastuzumab in terms of DFS. (Stage II) IV. To compare the sequential schedule of the combination of AC, weekly paclitaxel, and trastuzumab with the combination of AC followed by the combination of weekly paclitaxel and trastuzumab in terms of DFS. (Stage II) V. To compare the combination AC followed by weekly paclitaxel with the sequential schedule of the combination of AC, weekly paclitaxel, and trastuzumab in terms of the rate of cardiac events. (Stage II)

SECONDARY OBJECTIVES:

I. To compare the combination of AC followed by weekly paclitaxel with the sequential schedule of the combination of AC, weekly paclitaxel, and trastuzumab in terms of overall survival (OS).

II. To compare the combination AC followed by weekly paclitaxel with the combination of AC followed by the combination of weekly paclitaxel and trastuzumab in terms of OS.

III. To compare the sequential schedule of the combination AC, weekly paclitaxel, and trastuzumab with the combination of AC followed by the combination of weekly paclitaxel and trastuzumab in terms of OS.

TERTIARY OBJECTIVES:

I. To determine whether higher levels of shed ECD (extracellular domain) or autoantibodies to human epidermal growth factor receptor (HER)-2 and HER-1 measured in the serum prior to treatment are prognostic for DFS and survival.

II. To determine the concordance of central review of HER-2 overexpression as measured by the HercepTest (DAKO) and Vysis fluorescence in situ hybridization (FISH).

III. For each treatment arm, levels of brain natriuretic peptide (BNP), troponin-T (TnT), troponin-I (cTnI), tumor necrosis factor alpha (TNF-alpha), interleukin-1 beta (IL-1beta) and interleukin-6 (IL-6), CD40 ligand, and troponin levels will be compared and contrasted.

IV. To determine whether genetic markers are prognostic for cardiac adverse events associated with treatment.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I*: Patients receive doxorubicin hydrochloride intravenously (IV) and cyclophosphamide IV over 20-30 minutes on day 1. Treatment repeats every 3 weeks for 4 courses. Patients then receive paclitaxel IV over 1 hour beginning on day 1 of week 13 and continuing weekly for 12 courses in the absence of disease progression or unacceptable toxicity. NOTE: *Patients who completed paclitaxel on or after October 25, 2004 may receive trastuzumab for a maximum of 52 weeks either concurrently with paclitaxel or following completion of paclitaxel treatment.

ARM II*: Patients receive doxorubicin hydrochloride, cyclophosphamide, and paclitaxel as in arm I. Patients then receive trastuzumab IV over 30-90 minutes beginning on day 1 of week 25 and continuing weekly for 52 courses in the absence of disease progression or unacceptable toxicity. NOTE: *Patients who completed paclitaxel on or after October 25, 2004 may receive trastuzumab for a maximum of 52 weeks either concurrently with paclitaxel or following completion of paclitaxel treatment.

ARM III: Patients receive doxorubicin hydrochloride and cyclophosphamide as in arm I. Patients then receive paclitaxel IV over 1 hour and trastuzumab IV over 30-90 minutes beginning on day 1 of week 13 and continuing weekly for 12 courses. Patients then receive trastuzumab IV over 30 minutes beginning on day 1 of week 25 and continuing weekly for 40 courses in the absence of disease progression or unacceptable toxicity.

Within 5 weeks after completion of paclitaxel, patients may undergo radiotherapy. All postmenopausal estrogen receptor (ER)- or progesterone receptor (PR)-positive patients receive oral tamoxifen or an aromatase inhibitor once daily for 5 years beginning no later than 5 weeks after the last dose of paclitaxel. Patients may also receive an aromatase inhibitor once daily for 5 years after 5 years of daily tamoxifen. Patients who receive tamoxifen once daily for less than 4.5 years may receive an aromatase inhibitor daily until they have received a total of 5 years of adjuvant hormonal therapy.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 6 months for 4 years, and then annually for 15 years or until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Required tumor parameters for node positive disease: NOTE: This study will continue to use the American Joint Committee on Cancer (AJCC) 5th edition for TNM classification and staging

  * Operable, histologically confirmed adenocarcinoma of the female breast and positive lymph nodes

    * Node positivity may be determined by either an axillary node dissection or a positive sentinel node finding by hematoxylin and eosin (H&E)

      * NOTE: Positive nodes refers to H&E visible nodal metastases; immunohistochemistry (IHC) positive only cells in lymph nodes will not be considered positive nodes
    * One or more positive lymph nodes whose tumors are T1-3, pN1-2, M0 are eligible
    * cN2 disease is not eligible
    * pN2 disease is eligible
    * One positive lymph node by sentinel node biopsy or at least 6 axillary nodes must be examined on axillary node dissection with at least one positive lymph node
    * Metaplastic carcinoma is eligible
  * ER/PgR determination
  * HER-2 positive (pre-entry requirement for registration)

    * FISH must show gene amplification OR
    * IHC assay must show a strong positive (3+) staining score

      * NOTE: ductal carcinoma in situ (DCIS) components should not be counted in the determination of degree of IHC staining or FISH amplification
* Required tumor parameters for high-risk node-negative disease; NOTE: This study will continue to use the AJCC 5th edition for TNM classification and staging

  * Operable, histologically confirmed adenocarcinoma of the female breast and negative lymph nodes

    * Node status may be determined by either axillary node dissection or sentinel node biopsy with H&E staining; to be considered node negative, either of the following must be true: 1) negative sentinel node biopsy or 2) no positive lymph nodes found among at least 6 axillary nodes examined on axillary node dissection
    * NOTE: IHC positive only cells in lymph nodes will not be considered positive nodes
    * Tumors > 2.0 cm (irrespective of hormonal receptor status) or > 1.0 cm if ER-negative and PR-negative disease
  * ER/PgR determination
  * HER-2 positive (pre-entry requirement for registration)

    * FISH must show gene amplification OR
    * IHC assay must show a strong positive (3+) staining score

      * NOTE: DCIS components should not be counted in the determination of degree of IHC staining or FISH amplification
* =< 84 days from mastectomy or =< 84 days from axillary dissection or sentinel node detection if the patient's most extensive breast surgery was a breast sparing procedure; (This timing is per a decision by the Breast Intergroup)
* Surgical resection margins. All tumor should be removed by either a modified radical mastectomy or a segmental mastectomy with axillary node dissection

  * Mastectomy: There will be no evidence of gross or microscopic tumor (invasive or DCIS) at the surgical resection margins noted in the final surgery or pathology reports; patients with close margins are eligible
  * Segmental mastectomy (lumpectomy): Margins must be clear of invasive cancer and DCIS
  * Axillary dissection or sentinel node dissection: There will be no gross residual adenopathy
* TAM therapy

  * May have received up to four weeks of TAM therapy, or any other hormonal agent, for this malignancy
  * May have received TAM or raloxifene for purposes of chemoprevention (e.g., Breast Cancer Prevention Trial) or for other indications (including previous breast cancer if lobular carcinoma in situ [LCIS]) but must be discontinued before registration on this study
  * May never have received TAM, raloxifene, or any other hormonal agent
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelets (PLT) >= 100,000/mm^3
* Total bilirubin =< 1.5 x upper normal limit (UNL)
* Aspartate aminotransferase (AST) =< 2.0 x UNL
* Left ventricular ejection fraction (LVEF) within institutional normal range; if LVEF is > 75%, the investigator should consider performing a second review of the multigated acquisition (MUGA)/echocardiogram or performing a repeat MUGA/echocardiogram prior to registration; such re-reviews or repeat MUGA/echocardiogram are not permitted after registration
* Willingness to discontinue sex hormonal therapy, e.g., birth control pills, ovarian hormonal replacement therapy, etc., prior to registration and while on study
* Willingness to discontinue any hormonal agent such as raloxifene (Evista) prior to registration and while on study
* Non-breast malignancies that have not recurred within the last 5 years and are deemed to be at low risk for recurrence

EXCEPTIONS: These non-breast malignancies are eligible even if diagnosed =< 5 years prior to registration:

* Squamous or basal cell carcinoma of the skin that has been effectively treated
* Carcinoma in situ of the cervix that has been treated by surgery only
* Lobular carcinoma in situ (LCIS) of the ipsilateral or contralateral breast treated by surgery and/or tamoxifen only

  * Patients undergoing breast conservation therapy (i.e., lumpectomy and axillary dissection) must have plans to receive radiation therapy to the breast +/- regional lymphatics following completion of the chemotherapy; for patients treated with mastectomy, the use of radiation therapy is required for 4 or more positive lymph nodes and must be started after completion of chemotherapy; the use of radiation therapy is at the discretion of the investigator for 0-3 positive lymph nodes but, if used, must be started after the completion of chemotherapy
  * Prior to registration, the physician must designate if it is planned for the patient to receive radiation therapy (for adjuvant radiation therapy post-mastectomy or, less commonly, post-conservative therapy but not primary breast radiation as part of breast conserving treatment)
  * Willing and able to sign an informed consent
  * Gene amplified by FISH or strong positivity (3+) by HercepTest on central review; Note: The patient registers based on community HER-2 testing using FISH or IHC, AC chemotherapy is initiated; the tumor block or slides must be received =< 2 weeks from time of registration to the North Central Cancer Treatment Group (NCCTG) Operations Office for central HER-2 testing

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, intrauterine device [IUD], surgical sterilization, or abstinence, etc.); hormonal birth control methods are not permitted
* Locally advanced tumors (classification T4) at diagnosis including tumors fixed to chest wall, peau d'orange, skin ulcerations/nodules, or clinical inflammatory changes (diffuse brawny cutaneous induration with an erysipeloid edge)
* Prior history of breast cancer, except LCIS
* Bilateral invasive carcinoma, either metachronous or synchronous (EXCEPTION: Patients diagnosed with unilateral invasive carcinoma and metachronous or synchronous DCIS of the contralateral breast treated with mastectomy are eligible)
* Prior chemotherapy, radiation therapy, immunotherapy, or biotherapy for breast cancer
* Active, unresolved infection
* Active cardiac disease

  * Any prior myocardial infarction
  * History of documented congestive heart failure (CHF)
  * Current use of digitalis or beta-blockers for CHF
  * Any prior history of arrhythmia or cardiac valvular disease requiring medications or clinically significant
  * Current use of medications for treatment of arrhythmias or angina pectoris
  * Current uncontrolled hypertension (diastolic > 100 mmHg or systolic > 200 mmHg)
  * Clinically significant pericardial effusion
* Prior anthracycline or taxane therapy for any malignancy
* Sensitivity to benzyl alcohol
* Neurology/Neuropathy-Sensory >= grade 2 per the National Cancer Institute's (NCI's) Common Toxicity Criteria Version 2.0; EXCEPTION: Any chronic neurologic disorder will be looked at on a case-by-case basis by the study chair

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3436 (Actual)
Dates: Start 2000-05-19 (Actual); Primary Completion 2005-04-25 (Actual); Study Completion 2010-01-27 (Actual)

PRIMARY OUTCOMES:
Duration of DFS | Time from registration to first adverse event, assessed up to 15 years
  Will be estimated using the Kaplan-Meier method. A stratified log-rank test will be used to assess whether DFS differs with respect to the addition of trastuzumab to a chemotherapy regimen including AC and paclitaxel. Ninety-five percent confidence intervals will be reported for relative risks, for DFS at the 5-year point, and for absolute benefit as defined by differences in DFS and OS.

SECONDARY OUTCOMES:
Overall survival | Time from registration to death due to any cause, assessed up to 15 years
  Will be estimated using the Kaplan-Meier method. A stratified log-rank test will be used to assess whether OS differs with respect to the addition of trastuzumab to a chemotherapy regimen including AC and paclitaxel. Ninety-five percent confidence intervals will be reported for relative risks, for OS at the 5-year point, and for absolute benefit as defined by differences in DFS and OS.

CONTACTS AND LOCATIONS:
Overall Officials: Edith A Perez, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (157):
- United States (154):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Western Regional CCOP, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Community Cancer Institute, Clovis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Washington Hospital, Fremont, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - University of California San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - The Angeles Clinic and Research Institute - Santa Monica Office, Santa Monica, California
  - Santa Rosa Memorial Hospital, Santa Rosa, California
  - University of Colorado Hospital, Aurora, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Milford Regional Medical Center, Milford, Massachusetts
  - Saint Vincent Hospital/Reliant Medical Group, Worcester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Essentia Health Cancer Center, Duluth, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Washington University - Jewish, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Montana Cancer Consortium NCORP, Billings, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Oregon, Eugene, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Roper Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford NCI Community Oncology Research Program of the North Central Plains, Sioux Falls, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Sentara Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Saskatoon Cancer Centre, Saskatoon, Saskatchewan, Canada
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- University Of Pretoria, Pretoria, South Africa

REFERENCES:
- [Derived] Chumsri S, Pai T, Ma Y, Li Z, Gil A, Moreno-Aspitia A, Colon-Otero G, Pogue-Geile KL, Rasgoti P, Paik S, Perez EA, Thompson EA. Clinical Treatment Score Post-5 Years (CTS5) and Late Recurrence Risk in Hormone Receptor-Positive, HER2-Positive Breast Cancer. J Natl Compr Canc Netw. 2024 Aug 26;22(7):463-468. doi: 10.6004/jnccn.2024.7015. PMID 39191270
- [Derived] Chumsri S, Li Z, Serie DJ, Norton N, Mashadi-Hossein A, Tenner K, Brauer HA, Warren S, Danaher P, Colon-Otero G, Partridge AH, Carey LA, Hilbers F, Van Dooren V, Holmes E, Di Cosimo S, Werner O, Huober JB, Dueck AC, Sotiriou C, Saura C, Moreno-Aspitia A, Knutson KL, Perez EA, Thompson EA. Adaptive immune signature in HER2-positive breast cancer in NCCTG (Alliance) N9831 and NeoALTTO trials. NPJ Breast Cancer. 2022 May 24;8(1):68. doi: 10.1038/s41523-022-00430-0. PMID 35610260
- [Derived] Caparica R, Ma Y, De Angelis C, Richard F, Desmedt C, Awada A, Piccart M, Perez EA, Moreno-Aspitia A, Badve S, Thompson EA, de Azambuja E. Beta-2 Adrenergic Receptor Gene Expression in HER2-Positive Early-Stage Breast Cancer Patients: A Post-hoc Analysis of the NCCTG-N9831 (Alliance) Trial. Clin Breast Cancer. 2022 Jun;22(4):308-318. doi: 10.1016/j.clbc.2021.11.012. Epub 2021 Dec 2. PMID 34980541
- [Derived] Chumsri S, Li Z, Serie DJ, Mashadi-Hossein A, Colon-Otero G, Song N, Pogue-Geile KL, Gavin PG, Paik S, Moreno-Aspitia A, Perez EA, Thompson EA. Incidence of Late Relapses in Patients With HER2-Positive Breast Cancer Receiving Adjuvant Trastuzumab: Combined Analysis of NCCTG N9831 (Alliance) and NRG Oncology/NSABP B-31. J Clin Oncol. 2019 Dec 10;37(35):3425-3435. doi: 10.1200/JCO.19.00443. Epub 2019 Oct 17. PMID 31622131
- [Derived] Chumsri S, Serie DJ, Li Z, Pogue-Geile KL, Soyano-Muller AE, Mashadi-Hossein A, Warren S, Lou Y, Colon-Otero G, Knutson KL, Perez EA, Moreno-Aspitia A, Thompson EA. Effects of Age and Immune Landscape on Outcome in HER2-Positive Breast Cancer in the NCCTG N9831 (Alliance) and NSABP B-31 (NRG) Trials. Clin Cancer Res. 2019 Jul 15;25(14):4422-4430. doi: 10.1158/1078-0432.CCR-18-2206. Epub 2019 Feb 26. PMID 30808774
- [Derived] Norton N, Fox N, McCarl CA, Tenner KS, Ballman K, Erskine CL, Necela BM, Northfelt D, Tan WW, Calfa C, Pegram M, Colon-Otero G, Perez EA, Clynes R, Knutson KL. Generation of HER2-specific antibody immunity during trastuzumab adjuvant therapy associates with reduced relapse in resected HER2 breast cancer. Breast Cancer Res. 2018 Jun 14;20(1):52. doi: 10.1186/s13058-018-0989-8. PMID 29898752
- [Derived] Perez EA, Ballman KV, Tenner KS, Thompson EA, Badve SS, Bailey H, Baehner FL. Association of Stromal Tumor-Infiltrating Lymphocytes With Recurrence-Free Survival in the N9831 Adjuvant Trial in Patients With Early-Stage HER2-Positive Breast Cancer. JAMA Oncol. 2016 Jan;2(1):56-64. doi: 10.1001/jamaoncol.2015.3239. PMID 26469139
- [Derived] Perez EA, Baehner FL, Butler SM, Thompson EA, Dueck AC, Jamshidian F, Cherbavaz D, Yoshizawa C, Shak S, Kaufman PA, Davidson NE, Gralow J, Asmann YW, Ballman KV. The relationship between quantitative human epidermal growth factor receptor 2 gene expression by the 21-gene reverse transcriptase polymerase chain reaction assay and adjuvant trastuzumab benefit in Alliance N9831. Breast Cancer Res. 2015 Oct 1;17(1):133. doi: 10.1186/s13058-015-0643-7. PMID 26429296
- [Derived] O'Sullivan CC, Bradbury I, Campbell C, Spielmann M, Perez EA, Joensuu H, Costantino JP, Delaloge S, Rastogi P, Zardavas D, Ballman KV, Holmes E, de Azambuja E, Piccart-Gebhart M, Zujewski JA, Gelber RD. Efficacy of Adjuvant Trastuzumab for Patients With Human Epidermal Growth Factor Receptor 2-Positive Early Breast Cancer and Tumors </= 2 cm: A Meta-Analysis of the Randomized Trastuzumab Trials. J Clin Oncol. 2015 Aug 20;33(24):2600-8. doi: 10.1200/JCO.2015.60.8620. Epub 2015 Jun 22. PMID 26101239
- [Derived] Perez EA, Thompson EA, Ballman KV, Anderson SK, Asmann YW, Kalari KR, Eckel-Passow JE, Dueck AC, Tenner KS, Jen J, Fan JB, Geiger XJ, McCullough AE, Chen B, Jenkins RB, Sledge GW, Winer EP, Gralow JR, Reinholz MM. Genomic analysis reveals that immune function genes are strongly linked to clinical outcome in the North Central Cancer Treatment Group n9831 Adjuvant Trastuzumab Trial. J Clin Oncol. 2015 Mar 1;33(7):701-8. doi: 10.1200/JCO.2014.57.6298. Epub 2015 Jan 20. PMID 25605861
- [Derived] Perez EA, Romond EH, Suman VJ, Jeong JH, Sledge G, Geyer CE Jr, Martino S, Rastogi P, Gralow J, Swain SM, Winer EP, Colon-Otero G, Davidson NE, Mamounas E, Zujewski JA, Wolmark N. Trastuzumab plus adjuvant chemotherapy for human epidermal growth factor receptor 2-positive breast cancer: planned joint analysis of overall survival from NSABP B-31 and NCCTG N9831. J Clin Oncol. 2014 Nov 20;32(33):3744-52. doi: 10.1200/JCO.2014.55.5730. Epub 2014 Oct 20. PMID 25332249
- [Derived] Perez EA, Suman VJ, Davidson NE, Gralow JR, Kaufman PA, Visscher DW, Chen B, Ingle JN, Dakhil SR, Zujewski J, Moreno-Aspitia A, Pisansky TM, Jenkins RB. Sequential versus concurrent trastuzumab in adjuvant chemotherapy for breast cancer. J Clin Oncol. 2011 Dec 1;29(34):4491-7. doi: 10.1200/JCO.2011.36.7045. Epub 2011 Oct 31. PMID 22042958
- [Derived] Romond EH, Perez EA, Bryant J, Suman VJ, Geyer CE Jr, Davidson NE, Tan-Chiu E, Martino S, Paik S, Kaufman PA, Swain SM, Pisansky TM, Fehrenbacher L, Kutteh LA, Vogel VG, Visscher DW, Yothers G, Jenkins RB, Brown AM, Dakhil SR, Mamounas EP, Lingle WL, Klein PM, Ingle JN, Wolmark N. Trastuzumab plus adjuvant chemotherapy for operable HER2-positive breast cancer. N Engl J Med. 2005 Oct 20;353(16):1673-84. doi: 10.1056/NEJMoa052122. PMID 16236738